CLINICAL TRIAL: NCT00264342
Title: Safety of Nicotine Reduction Strategy
Brief Title: Effectiveness of Using Reduced Nicotine Cigarettes in Men and Women Smokers to Combat Nicotine Addiction
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: R01CA078603-05A1 (NIH)
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Nicotine Dependence; Tobacco Use Disorder
Keywords: Smoking; Tobacco; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue (blood) and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a 2-year study involving the progressive reduction in the nicotine content of cigarettes. The investigators believe that at the end of the study smokers of cigarettes with progressively reduced nicotine content will be "weaned" from nicotine. At the end of the study, the result will be a decreased level of nicotine dependence. When smokers are again free to choose any smoking behavior, they will smoke fewer cigarettes and/or have a greater interest in quitting compared to a control group that smokes their usual cigarettes.

DETAILED DESCRIPTION:
This is a 2-year, randomized, two-arm study involving a 6-month period of progressive reduction in the nicotine content of cigarettes. During the first year (tapering/maintenance phases), subjects will smoke progressively reduced nicotine content (RNC) cigarettes over a period of six months, and then remain on the lowest nicotine content cigarette for an additional six months. Comparisons will be made with a control group in which subjects will smoke their usual normal nicotine yield cigarettes. There will be a one year follow-up phase during which subjects will be monitored and will be free to resume smoking a commercial cigarette of their choice, or to quit.

We hypothesize that smokers of cigarettes with progressively reduced nicotine content will experience a reduction in nicotine intake without compensatory oversmoking. This will serve to "wean" them from nicotine and result in a decreased level of nicotine dependence. Once this has occurred, subjects will then be able to maintain their reduced level of nicotine intake for the 6 months that they continue smoking the lowest level RNC cigarette. When they are again free to choose any smoking behavior (follow-up phase), as a result of the period of lowered dependence they will smoke fewer cigarettes and/or have a greater interest in quitting compared to the control group, whose level of nicotine dependence is hypothesized to be sustained throughout.

Primary Hypotheses:

1. Nicotine intake will be lower for the RNC group than for the control group.
2. Exposure to tobacco smoke gas phase constituents will be similar for the RNC and control group.
3. Exposure to tobacco smoke tar constituents will be similar for the RNC and control group.
4. Cardiovascular biomarkers of inflammation, platelet activation, endothelial dysfunction, and HDL cholesterol will be lower for the RNC group than for the control group.
5. Cigarette consumption, as measured by cigarettes-per-day (CPD), will be lower for the RNC group than for the control group.

Secondary hypotheses:

1. Over the course of tapering and maintenance and at follow-up, interest in quitting will be higher in the RNC group compared to the control group.
2. At follow-up, measures of cigarette consumption, nicotine intake, and exposure to tobacco smoke combustion constituents will be lower for the RNC group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and screening blood tests
* Current moderate-to-heavy smoker as determined by:

  1. smoking more than 10 cigarettes per day regularly for the past year (by history); and
  2. expired carbon monoxide (CO) at screening visit of 25 ppm or more and/or plasma cotinine level of 100 ng/ml or more.
* Age 18-70 years
* Any racial/ethnic background

Exclusion Criteria:

* Expressed desire to quit smoking within 6 months.
* Significant medical conditions (such as anemia, heart disease, uncontrolled hypertension, thyroid disease, diabetes, renal or liver impairment, glaucoma, or prostatic hypertrophy) or psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder, or current regular use of psychiatric medications such as major tranquilizers and antidepressants). Smokers with uncomplicated controlled hypertension may be enrolled.
* Pregnancy or lactation (by history)
* Current use of smokeless tobacco, pipes or cigars
* Alcohol abuse or illicit drug use (by history)
* Concurrent participation in another clinical trial or prior participation in our pilot studies using the same RNC cigarettes as in these studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adults 18 and over
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2005-07; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Benowitz NL, Jacob P 3rd, Bernert JT, Wilson M, Wang L, Allen F, Dempsey D. Carcinogen exposure during short-term switching from regular to "light" cigarettes. Cancer Epidemiol Biomarkers Prev. 2005 Jun;14(6):1376-83. doi: 10.1158/1055-9965.EPI-04-0667. PMID 15941944
- [Background] Gray N, Henningfield JE, Benowitz NL, Connolly GN, Dresler C, Fagerstrom K, Jarvis MJ, Boyle P. Toward a comprehensive long term nicotine policy. Tob Control. 2005 Jun;14(3):161-5. doi: 10.1136/tc.2004.010272. PMID 15923465
- [Background] Hukkanen J, Jacob P 3rd, Benowitz NL. Metabolism and disposition kinetics of nicotine. Pharmacol Rev. 2005 Mar;57(1):79-115. doi: 10.1124/pr.57.1.3. PMID 15734728
- [Background] Arcavi L, Benowitz NL. Cigarette smoking and infection. Arch Intern Med. 2004 Nov 8;164(20):2206-16. doi: 10.1001/archinte.164.20.2206. PMID 15534156
- [Background] Swan GE, Benowitz NL, Jacob P 3rd, Lessov CN, Tyndale RF, Wilhelmsen K, Krasnow RE, McElroy MR, Moore SE, Wambach M. Pharmacogenetics of nicotine metabolism in twins: methods and procedures. Twin Res. 2004 Oct;7(5):435-48. doi: 10.1375/1369052042335269. PMID 15527659
- [Derived] Benowitz NL, Gan Q, Goniewicz ML, Lu W, Xu J, Li X, Jacob P 3rd, Glantz S. Different profiles of carcinogen exposure in Chinese compared with US cigarette smokers. Tob Control. 2015 Dec;24(e4):e258-63. doi: 10.1136/tobaccocontrol-2014-051945. Epub 2014 Dec 22. PMID 25535294
- See also: UCSF Nicotine and Tobacco Research — http://tobacco.ucsf.edu